CLINICAL TRIAL: NCT03041168
Title: Evaluation of a Novel Technique to Investigate CAS Piezo Electric Sensors
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to suspension of funding from CVR Global.
Sponsor: Thomas Jefferson University (Other)
Collaborators: CVR Global, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16G.774
Record Dates: First submitted 2017-01-11; First posted 2017-02-02 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Carotid Stenotic Scan — Each subject will have been scheduled for a carotid ultrasound, or other imaging test of the neck (carotids) as ordered by his/her physician for clinical or screening purposes. These studies will be read by a Jefferson radiologist and a report generated for standard clinical purposes. These reports and the images will be collected and de-identified to be used as comparator measurements to the CSS results. The CSS device is shaped like a stethoscope with 3 small gel pads. It is positioned with a gel pad on either side of the neck and one on the front of the chest. The scan takes about 1-2 minutes to provide an image on the screen of the device cart. The scan device pads just lie on the skin and do not use any invasive techniques to provide the image.

SUMMARY:
The proposed study is evaluating a novel technology, Carotid Stenotic Scan (CSS), developed by the sponsor, CVR Global. Study Design. This is a prospective cohort study that will compare a new application of a technology, the CSS device, to reference standards for assessment of carotid disease.

DETAILED DESCRIPTION:
The overall objectives of this study are to demonstrate that the Carotid Stenotic Scan (CSS) can accurately detect significant carotid artery stenosis.

Secondary objective is to relate changes in CSS signal to different degrees of stenosis. We obtain a "proof of concept" if the device correlates strongly with the established classification of atherosclerotic carotid disease derived various imaging modalities including magnetic resonance angiography (MRA) and computer tomographic angiography (CTA), conventional angiography, or carotid ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 referred for carotid duplex ultrasound.
* Subjects over 18 referred for CT angiography, MR angiography, or conventional angiography of the carotid arteries

Exclusion Criteria:

* Previous history of carotid endarterectomy, carotid artery stent
* Previous surgery involving the neck (including thyroidectomy or parathyroidectomy)
* Patients with prosthetic heart valve
* Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients presenting to a Jefferson facility for carotid imaging studies. Subjects scheduled for carotid artery assessments will be identified prior to the day of study using radiology scheduling.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2017-01; Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Difference between percent carotid artery stenosis measured by CSS and by carotid ultrasound | CSS reported percentage of carotid stenosis within 30 days of carotid ultrasound

SECONDARY OUTCOMES:
Difference between percent carotid artery stenosis measured by CSS and by carotid CTA | CSS reported percentage of carotid stenosis within 30 days of carotid CTA
Difference between percent carotid artery stenosis measured by CSS and by carotid MRA | CSS reported percentage of carotid stenosis within 30 days of carotid MRA
Difference between percent carotid artery stenosis measured by CSS and carotid angiogram | CSS reported percentage of carotid stenosis within 30 days of carotid angiogram

CONTACTS AND LOCATIONS:
Overall Officials: David J Whellan, MD MHS, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No